CLINICAL TRIAL: NCT03775993
Title: Treatment of Growth Hormone Deficiency Associated With Chronic Heart Failure: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Treatment of GHD Associated With CHF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-004580-39
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Growth Hormone Deficiency
Keywords: Growth Hormone; Placebo; Exercise capacity; Vascular reactivity; LV function; Prognosis
MeSH Terms: conditions — Heart Failure; Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GHD (Active Comparator)
  Interventions: Drug: Human growth hormone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Human growth hormone — Administration of growth hormone
  Arms: GHD
Other: Placebo — Administration of placebo
  Arms: Placebo

SUMMARY:
Aim of the current study is to assess the cardiovascular effects of GH replacement therapy in patients with coexisting GHD and CHF

DETAILED DESCRIPTION:
Multiple anabolic deficiencies are common in chronic heart failure (CHF) and identify subgroups of patients with higher mortality. Apart from CHF, GH deficiency (GHD) per se increases cardiovascular mortality in the general population and low IGF-1 levels in the general population predict the development of ischemic heart disease and CHF. GHD modifies cardiac size and function, through a reduction in both myocardial growth and cardiac performance. The investigators therefore completed 2 studies aimed at evaluating the clinical status, neurohormonal parameters, exercise capacity, vascular reactivity, and left ventricular architecture and function in patients with GHD and CHF, at baseline and after 6 months of GH replacement therapy. They subsequently extended the observation period up to 48 months. At 6-months, GH replacement therapy improved clinical status and exercise capacity, as shown by a significant reduction of the Minnesota living with heart failure questionnaire score, increased peak oxygen consumption and exercise duration, and flow mediated vasodilation of the brachial artery. No major adverse events were reported in the patients receiving GH.

However, the encouraging results of these studies are limited by the lack of a double-blind, placebo-controlled design, insofar as the investigators performed a randomized controlled, single-blind study.

ELIGIBILITY:
Inclusion Criteria:

1. patients of either sex affected by CHF NYHA class I-III, secondary to ischemic or idiopathic di-lated cardiomyopathy;
2. age range 18-85 years;
3. stable and optimal medical therapy for at least three months prior to randomization, including ACE inhibitors or AT1 antagonists and beta-blockers (unless untolerated);
4. LV ejection fraction 40% or less and LV end-diastolic dimension 55 mm or more;
5. GH deficiency diagnosed with GHRH + arginine provocative test;
6. signed informed consent.

Exclusion Criteria:

1. inability to perform a bicycle exercise test;
2. poorly controlled diabetes mellitus (HbA1c >8.5) and/or active proliferative or severe non-proliferative diabetic retinopathy;
3. active and/or history of malignancy;
4. unstable angina or recent myocardial infarction (less than six months);
5. severe liver or kidney disease (serum creatinine levels >2.5 mg/dl

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of peak oxygen consumption (peak VO2) | 1 year
  According to previous observations, the investigators set a target increase of peak VO2 in the treated arm at 3 ml/kg/min at the end of the study

SECONDARY OUTCOMES:
Number of Hospitalizations | 1 year
End-systolic LV volumes | 1 year
NT-proBNP levels | 1 year
Quality of life score from the Minnesota Living with Heart Failure Questionnaire | 1 year
  The questionnaire is comprised of 21 physical, emotional and socioeconomic questions that may adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (lower valure) to 5 (upper value) scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The final score is calculated by sum.
Evaluation of Endothelial function (flow-mediated vasodilation) | 1 year
Muscle strength (handgrip) | 1 year
Evaluation of the Levels of Endothelial Progenitor Cells (EPCs) | 1 year
Evaluation of the Levels of lymphocyte G protein-coupled receptor kinase (GRK)-2 | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marra AM, D'Assante R, De Luca M, Arcopinto M, Gargiulo P, Valente V, Crisci G, Rainone C, Modestino M, Giardino F, Paolillo S, Cacciatore F, Saldamarco L, Bruzzese D, Scarpa D, Filardi PP, Esposito G, Sacca L, Bossone E, Salzano A, Cittadini A. Growth Hormone Replacement Therapy in Heart Failure With Reduced Ejection Fraction: A Randomized, Double-Blind, Placebo-Controlled Trial. JACC Heart Fail. 2025 Apr;13(4):602-614. doi: 10.1016/j.jchf.2024.11.017. Epub 2025 Mar 5. PMID 40047762